CLINICAL TRIAL: NCT00518765
Title: A Single-center, Placebo-controlled Study of the Effects of Ascending Single Oral Doses of Aliskiren Compared With Captopril on Renal Hemodynamics in Healthy Volunteers on a Low and High Sodium Diet "Renin Inhibition and the Kidney"
Brief Title: Hemodynamic Effects of Aliskiren Compared to Captopril on the Kidney in Healthy Volunteers on a Low- and High- Sodium Diet
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CSPP100A2318
Expanded Access: Available
Record Dates: First submitted 2007-08-20; First posted 2007-08-21 (Estimated); Last update posted 2010-10-06 (Estimated); Status verified 2010-10

CONDITIONS: Hypertension
Keywords: aliskiren, renal hemodynamics, hormonal response, renin pathway, RAAS biomarkers
MeSH Terms: conditions — Hypertension | interventions — aliskiren

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Various sequences of different doses of Aliskiren
  Interventions: Drug: Aliskiren
- 2 (Experimental): Various sequences of different doses of Aliskiren plus placebo
  Interventions: Drug: Aliskiren plus placebo
- 3 (Experimental): Various sequences of different doses of Aliskiren
  Interventions: Drug: Aliskiren
- 4 (Experimental): Various sequences of different doses of Aliskiren plus placebo
  Interventions: Drug: Aliskiren plus placebo

INTERVENTIONS:
Drug: Aliskiren
  Other Names: SPP100
  Arms: 1
Drug: Aliskiren plus placebo
  Arms: 2
Drug: Aliskiren
  Other Names: SPP100
  Arms: 3
Drug: Aliskiren plus placebo
  Arms: 4

SUMMARY:
This study will measure the effects of different doses of aliskiren on kidney blood flow and function in healthy adults and determine how salt intake affects the response to aliskiren.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects age 18 to 75 years of age included
* Strictly adhere to provided diet.

Exclusion Criteria:

* Symptomatic low blood pressure
* Prescription medications, including those for blood pressure control, birth control pills, and any other medication that could affect kidney function
* Over-the-counter medication 2 weeks before study start
* Clinically significant heart abnormalities.
* Previous history of allergy to the study drug or drugs similar to the study drug.
* Any surgical or medical condition which might significantly alter the action of a drug (for example, absorption, distribution, metabolism or excretion) or which may jeopardize the subject in case of participation in the study.

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-10; Primary Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Renal plasma flow following 3 single doses of aliskiren in healthy volunteers on a low sodium(10 mEq/day)diet | baseline and hourly intervals.

SECONDARY OUTCOMES:
Single dose application of aliskiren on renal hemodynamics and circulating markers of the renin pathway | baseline, and at 5 hours, and 24 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigative site
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Fisher ND, Jan Danser AH, Nussberger J, Dole WP, Hollenberg NK. Renal and hormonal responses to direct renin inhibition with aliskiren in healthy humans. Circulation. 2008 Jun 24;117(25):3199-205. doi: 10.1161/CIRCULATIONAHA.108.767202. Epub 2008 Jun 16. PMID 18559696